CLINICAL TRIAL: NCT04958161
Title: Reconditioning Exercise for COVID-19 Patients Experiencing Residual sYmptoms
Acronym: RECOVERY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll anyone.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00075690
Record Dates: First submitted 2021-07-08; First posted 2021-07-12 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: exercise; rehabilitation; physical function
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Therapy (Experimental): Exercise therapy will be performed three times per week for 12 weeks.
  Interventions: Other: Exercise Therapy
- Wait List Control (No Intervention): Wait-list-control participants will be asked to continue their normal activities over the 12 week period.

INTERVENTIONS:
Other: Exercise Therapy — Each exercise session will involve 5 to10 minutes of stretching and slow walking followed by a 30 minute stimulus phase of aerobic exercise. Exercise intensity during the stimulus phase will be prescribed based on the graded exercise test results and will be gradually increased with the goal of the participant exercising continuously for 30 minutes at 50% to 85% of symptom-limited maximum heart rate, or maintained at a level below that which causes symptomatic or silent ischemia. Following the aerobic phase of exercise, participants will complete one set of 8 to 12 repetitions of muscle-strengthening activities for all major muscle groups (legs, hips, back, abdomen, chest, shoulders, and arms). Participants will be provided with a home based aerobic exercise program. They will be encouraged to perform this home-based program twice a week on days when they are not attending the center-based program.
  Arms: Exercise Therapy

SUMMARY:
Individuals who had COVID-19 and are thought to have recovered from the disease often experience long-term symptoms such as fatigue, extreme tiredness and shortness of breath, a condition referred to as Long COVID. Previous studies have shown that regular exercise is beneficial for individuals suffering similar symptoms as a result of other diseases such as Chronic Fatigue Syndrome. The goal of this study is determine if participation in a three-month structured exercise program will improve physical function in individuals suffering from Long COVID.

DETAILED DESCRIPTION:
In December of 2019, a previously unknown betacoronavirus was discovered in the airways of patients with pneumonia in Wuhan, China. The novel coronavirus disease (COVID-19) caused by the virus (severe acute respiratory syndrome coronavirus (SARS-CoV-2)) spread rapidly around the world. Common symptoms include cough, fever, dyspnea (i.e. shortness of breath), musculoskeletal aches and pains and fatigue. These symptoms, most notably fatigue and dyspnea, have been reported months after the onset of the disease and often long after patients are thought to have recovered from the disease. Between one and two thirds of patients with milder forms of the disease report symptoms up to two months after the onset of symptoms. This condition is now referred to as Long COVID or Post- Acute Sequelae of SARS-CoV-2 infection, and the characteristic symptoms of this condition are dyspnea and extreme fatigue. Additionally, pulmonary, musculoskeletal, neurological, cardiac, and psychological sequelae in these survivors can affect their physical function and ability to perform activities of daily living. While exercise rehabilitation in patients recovering from COVID-19 has been cautiously recommended, there is little known about the response to exercise in patients with Long COVID-19 nor the optimal methods or strategies for rehabilitating these patients. Understanding the responses to an exercise program is instrumental in designing safe and effective rehabilitation strategies for these patients. The objective of this study is to examine the effect of a 3-month exercise therapy program on physical function in individuals who have recovered from COVID-19 between the previous 2 to 6 months, yet still report symptoms of the disease. The study is a randomized, wait-list-control pilot study designed to gather preliminary data. Participants will be randomized into one of two groups: an immediate treatment group or a wait-list-control group. The immediate treatment group will begin the exercise therapy program following randomization and will participate in the exercise program for a duration of three months. The wait-list-control group will receive usual care for the first three months, after which they will be allowed the opportunity to participate in the exercise therapy program for three months. Outcome measures will me made prior to randomization and following either the three-month exercise program or three months of usual care.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Able to read and speak English
* Proof of a positive nucleic acid amplification test for the determination of COVID-19
* Two months post positive nucleic acid amplification test for the determination of COVID
* Self-report of COVID-19 symptoms (symptoms include any of the following: reduced exercise capacity, fatigue, cough, shortness of breath, headache and/or joint pain)
* Able to understand and willing to sign a written informed consent document
* Willing and able to complete all study procedures including attending all exercise sessions

Exclusion Criteria:

* Currently exercising more than 60 minutes per week at a moderate intensity or 30 minutes per week at a high intensity
* Current use of supplemental oxygen
* Active treatment for cancer
* Severe congestive heart failure, pulmonary disease, stroke, peripheral vascular disease, coronary artery disease and/or valvular heart disease
* Positive graded exercise test
* Major psychiatric disease
* Severe liver or hepatic disease
* Uncontrolled hypertension or diabetes
* Orthopedic impairment that prevents participation in an exercise program
* Blindness
* BMI > 40kg/m2
* Living more than 35 miles from exercise facility
* Plans to move within the next 6 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Performance Based Physical Function | Baseline
  Six minute walk distance will be used to measure performance based physical function. Subjects will walk at their chosen pace for six minutes on a pre-determined course. Total distance walked will be recorded.
Performance Based Physical Function | Week 12
  Six minute walk distance will be used to measure performance based physical function. Subjects will walk at their chosen pace for six minutes on a pre-determined course. Total distance walked will be recorded.
Self-reported Physical Function | Baseline
  The Physical Functioning scale of the Medical Outcomes 36 Item Short Form (SF-36) will be used to measure self-reported physical function. Patient responses are rated on a on a 3-point scale (1- yes, limited a lot; 2 - yes, limited a little; or 3- no, not limited at all) and will then be normalized with a mean of 50 and standard deviation of 10.
Self-reported Physical Function | Week 12
  The Physical Functioning scale of the Medical Outcomes 36 Item Short Form (SF-36) will be used to measure self-reported physical function. Patient responses are rated on a on a 3-point scale (1- yes, limited a lot; 2 - yes, limited a little; or 3- no, not limited at all) and will then be normalized with a mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
Physical Function | Baseline and Week 12
  Physical functioning will also be assessed using the Short Physical Performance Battery (SPPB). The SPPB score is based on timed measures of standing balance, walking speed, and ability to rise from a chair. Scores on each measure range from 0 - 4 and will be summed for a final score. Scores for the SPPB range from 0 to 12 with higher scores indicative of greater physical function.

OTHER OUTCOMES:
Lung Volumes and Capacities | Baseline and Week 12
  Nitrogen (N2) washout will be used to measure the various lung volumes and lung capacities according to American Thoracic Society and European Respiratory Society guidelines.
Air Flow | Baseline and Week 12
  Air flow out of the lungs will be measured using spirometry. The forced expiratory volume in one second (FEV1) will be measured according to American Thoracic Society and European Respiratory Society guidelines.
Diffusion Capacity | Baseline and Week 12
  Gas exchange will be used to measure the diffusion capacity of the lungs. All measures will be made according to American Thoracic Society and European Respiratory Society guidelines.
Respiratory Muscle Weakness | Baseline and Week 12
  Maximum inspiratory strength and maximum expiratory strength will be used to determine respiratory muscle weakness. Maximum inspiratory strength and maximum expiratory strength will be measured as pressures at the mouth generated at residual volume and total lung capacity, respectively. All measures will be made according to American Thoracic Society and European Respiratory Society guidelines.
Exercise Capacity | Baseline and Week 12
  Peak oxygen consumption (ml/kg/min) or aerobic capacity will be measured directly during a graded exercise test on an electronically braked cycle ergometer.
Cognitive Function | Baseline and Week 12
  The Montreal Cognitive Assessment (MoCA) will be used to characterize global cognitive function. Scores range from 0 to 30, with a score of 26 and higher considered normal.
Generic Health Related Quality of Life (HRQL) - Physical Component | Baseline and Week 12
  The SF-36 will be used as a generic measure of HRQL. The SF-36 consists of eight scales. Four of the eight scales will be used to produce a Physical Component score ranging from 0 -100 with lower scores indicative of poorer physical health.
Generic Health Related Quality of Life (HRQL) - Mental Component | Baseline and Week 12
  The SF-36 will be used as a generic measure of HRQL. The SF-36 consists of eight scales. Four of the eight scales will be used to produce a Mental Component score ranging from 0 -100 score with lower scores indicative of poorer mental health.
Disease Specific Health Related Quality of Life (HRQL) | Baseline and Week 12
  St. George's Respiratory Questionnaire (SGRQ) will be used as a disease specific measure of HRQL. SGRQ consists of three sub-scales. All three scales will be used to produce a score ranging from 0 - 100 score with lower scores indicative of a poorer health related quality of life.
Disability | Baseline and Week 12
  The Functional Performance Inventory - Short Form (FPI-SF) will be used to assess disability. The FPI-SF queries participants about performance of activities of daily living to assess disability. Scores range from 0 to 3 with higher scores reflecting better functioning.
Fatigue | Baseline and Week 12
  The Chalder Fatigue Score (CFQ-11) will be used to measure the severity of fatigue. Scores range from 0 to 33. Persons without fatigue problems would score 11 or lower.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Berry, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
Access Criteria: IPD that underlie results in a publication will be posted to a publicly accessible website following publication.